CLINICAL TRIAL: NCT05065307
Title: Effect of the Format of a Video Game on Children's Experience During Venipuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Cyril Sahyoun, Deputy Chief, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-00979
Record Dates: First submitted 2021-08-13; First posted 2021-10-04 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Pain, Procedural
Keywords: Hypnosis; Virtual Reality; Behavioral intervention; Venipuncture
MeSH Terms: conditions — Pain, Procedural | interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video game in Virtual reality (Experimental): The study subject will be playing a video game during the venipuncture, in virtual reality
  Interventions: Diagnostic Test: Venipuncture
- Video game on a tablet (Active Comparator): The study subject will be playing a video game during the venipuncture, on a tablet
  Interventions: Diagnostic Test: Venipuncture

INTERVENTIONS:
Diagnostic Test: Venipuncture — Diagnostic venipuncture

SUMMARY:
Anxiolysis and analgesia are of paramount importance when conducting medical procedures, particularly in children. Nonpharmacologic techniques such as distraction and hypnosis improve the patient experience when used in the correct setting and may reduce the need for medications and pharmacological sedation. Virtual reality immersion is a novel approach to anxiolysis and analgesia but the content (i.e. games) available on the market are limited in their appropriateness for age, and the lack of specific design for medical procedures. VRelief, designed using a multidisciplinary team of clinicians, hypnosis practitioners, psychologists and computer scientists specializing in the Multimodal Modelling of Emotion & Feeling may present a safe and superior alternative to a similar game presented in a video tablet format, in mitigating procedural anxiety and pain and improving the patient experience during venipuncture.

DETAILED DESCRIPTION:
Pain and anxiety experienced in the acute care setting remain a major global problem, resulting in high costs for those involved as well as for health care institutions. Pain and anxiety management techniques affect the quality of the care experienced by patients, relatives, and healthcare workers. Pharmacological procedures remain the most widely used approach, although they have important limitations, such as potential for adverse effects and dosing errors, especially in the most vulnerable populations such as young children. Non-pharmacological approaches to analgesia and anxiolysis have been explored, among which placebo, expectant, distraction, positive induction, reward, self-regulation, relaxation and hypnosis. Unfortunately, translational applications have been only partially successful, due to the limited and variable effectiveness of each approach, which often requires active and continuous patient cooperation. Hypnosis is an effective but incomplete approach that requires the presence of a specialist and can only be practiced from a certain age.

Virtual Reality (VR) is a promising technology that combines all of these methods above into an immersive and engaging tool for pain and anxiety relief that could equal or exceed the effectiveness of other existing non-pharmacological techniques. In addition, it is relatively inexpensive and provides a relevant alternative when hypnosis practitioners are not available.

The virtual reality contents (hereon ''games'') available on the market are varied. However, these tools are mainly based on distraction and often do not take into account the therapeutic communication and hypnosis principles proven useful in managing anxious children, as well as other psychological factors facilitating, for example, the "empowerment" of patients. Moreover, the quality of immersion in a virtual environment is essential for its effectiveness, and the tools currently available remain limited in this respect (mini-games, 360-degree video). Moreover, these tools have little external control and even fewer intelligent mechanisms to adapt content to the patient experience.

The investigators developed a prototype VR tool, which, unlike tools from other clinical studies of virtual reality, implemented a narration integrating several properties of hypnosis induction (in particular relaxation and regulation) with a gameplay designed to induce distraction and empowerment. The game was developed with the objective of engaging the child in an environment where he or she is first familiarized and reassured, then engaged in the missions of the game, and finally rewarded, all with the intent of decreasing anxiety and pain during a procedure. The investigators have carefully adapted the initial versions of this VR scenario to young, hospitalized children (starting from the age of 5 years of age) undergoing painful and anxiogenic procedures such as venipuncture. This population is ideal for our needs because they are often resistant to other non-pharmacological techniques (hypnosis susceptibility peaks between 8 and 12 years and, at the same time, have a good knowledge of artificial environments and computer games. A pilot study conducted in our department showed that children who played the VR game rated their pain and anxiety less high than children who received standard of care, during venipuncture. Venipuncture is some of the most common procedures in pediatric emergency departments and one of the most common sources of unrelieved pain and anxiety in hospitalized children.

To date, no study has attempted to isolate the added value of VR by comparing it with a similar game offered in a format such as a video tablet (ie.g.: iPad, etc.).

When used in a correct subset of patients (excluding patients with light-sensitive epilepsy), there are no risks anticipated aside from potential mild nausea or dizziness, which is rarely described in children using virtual reality, which would make this study a risk category A study.

ELIGIBILITY:
Inclusion Criteria:

- Children 5-12 undergoing a venipuncture as part of the Corona Immunitas Covid serology study

Exclusion Criteria:

* Parents prefer their child not to use screens
* Known or suspected light-sensitive epilepsy
* Moderate or severe intellectual disability
* Physical factors preventing placement of the VR headset (e.g.: wound on the face, etc.)
* Inability to understand or follow the procedures of the study due to a language barrie

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Child rating of maximum pain | during venipuncture
  Visual Analog Scale rating of minimum 0 (least amount) and maximum 10 (most amount)
Child rating of time spent thinking about pain | during venipuncture
  Visual Analog Scale rating of minimum 0 (least amount) and maximum 10 (most amount)
Child rating of anxiety | during venipuncture
  Visual Analog Scale rating of minimum 0 (least amount) and maximum 10 (most amount)
"Fun" rating | during venipuncture
  Visual Analog Scale rating of minimum 0 (least amount) and maximum 10 (most amount)
Parental rating of satisfaction | during venipuncture
  Visual Analog Scale rating of minimum 0 (least amount) and maximum 10 (most amount)

SECONDARY OUTCOMES:
Child rating of venipuncture unpleasantness | during venipuncture
  Visual Analog Scale rating of minimum 0 (least amount) and maximum 10 (most amount)
Heart rate change during the venipuncture compared to the start of the procedure | baseline, during the intervention, immediately after the intervention and 5 minutes later
  Visual Analog Scale rating of minimum 0 (least amount) and maximum 10 (most amount)
Number of persons required for physical and pharmacological restraint of children during these procedures | during venipuncture
  Visual Analog Scale rating of minimum 0 (least amount) and maximum 10 (most amount)
Feeling of immersion into the game | during venipuncture
  Visual Analog Scale rating of minimum 0 (least amount) and maximum 10 (most amount)
Parental anxiety | during venipuncture
  Visual Analog Scale rating of minimum 0 (least amount) and maximum 10 (most amount)
Healthcare worker rating of satisfaction | during venipuncture
  Visual Analog Scale rating of minimum 0 (least amount) and maximum 10 (most amount)

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Sahyoun, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Zavlanou C, Savary V, Mermet S, Sander D, Corradi-Dell'Acqua C, Rudrauf D, Tisserand Y, Sahyoun C. Virtual reality vs. tablet for procedural comfort using an identical game in children undergoing venipuncture: a randomized clinical trial. Front Pediatr. 2024 May 13;12:1378459. doi: 10.3389/fped.2024.1378459. eCollection 2024. PMID 38803637